CLINICAL TRIAL: NCT06277895
Title: Application of Emergency Rapid Detection of Expiratory Volatile Organic Compounds (VOCs) in Patients With Acute Cardiogenic Chest Pain
Brief Title: VOCs in Patients With Acute Cardiogenic Chest Pain
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Qilu Hospital of Shandong University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: KYLL-202401-047
Record Dates: First submitted 2024-01-25; First posted 2024-02-26 (Actual); Last update posted 2024-02-26 (Actual); Status verified 2024-01

CONDITIONS: Acute Coronary Syndrome; Acute Aortic Syndrome
MeSH Terms: conditions — Acute Coronary Syndrome; Acute Aortic Syndrome

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- cardiogenic chest pain group (Experimental): cardiogenic chest pain group/acute coronary syndrome
  Interventions: Diagnostic Test: VOCs
- normal group (Other): Healthy population
  Interventions: Diagnostic Test: VOCs

INTERVENTIONS:
Diagnostic Test: VOCs — test the end-expiratory gas

SUMMARY:
The goal of this observation study is to compare VOCs in cardiogenic chest pain population/health conditions, to answer：Establishment and promotion of the application system of emergency rapid detection of expiratory Volatile Organic Compounds (VOCs) in patients with acute cardiogenic chest pain

1. VOCs levels were measured at baseline in healthy people, and markers of VOCs that could be used to identify acute cardiogenic chest pain were sought.
2. The relationship between abnormal VOCs (mainly aldehydes) and prognosis of patients and the correlation with Super-score for early warning of acute heart failure.

ELIGIBILITY:
Inclusion Criteria:

Observation group inclusion criteria:

1. Over 18 years old, male or female;
2. Patients with acute cardiogenic chest pain (see diagnostic criteria);
3. Patient's informed consent.

Inclusion criteria of healthy control group:

1. Over 18 years old, male or female;
2. Centerless cerebrovascular disease, lung disease, no abnormal liver and kidney function, no acute infection recently;
3. Informed consent.

Exclusion Criteria:

1. The patient had difficulty in collecting breath;
2. Patients with terminal illness or receiving palliative care;
3. Have participated in other clinical studies or consider it inappropriate to participate in this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1400 (Estimated)
Dates: Start 2024-01-26 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Baseline VOCs (aldehydes) levels in healthy population | Baseline
  Baseline VOCs (aldehydes) levels in healthy population

SECONDARY OUTCOMES:
MACE in patients with cardiogenic chest pain | From enrollment to the end of treatment at 30 days
  the relationship between the different VOCs levels and 30-day MACE in patients with cardiogenic chest pain

CONTACTS AND LOCATIONS:
Locations (1):
- Qilu hospital, Jinan, Shandong, China